CLINICAL TRIAL: NCT05054075
Title: Methodological Design for Evaluating the Immune Capacity of Bivalve Fluids From Anodonta Cygnea in SARS and COVID-19 Human Infection: Intelligent Medicine Integration.
Brief Title: Protocol Design for Evaluating the Immunity of Bivalve Fluids From Anodonta Cygnea in SARS and COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade do Porto (Other)
Collaborators: Instituto Politécnico de Bragança (Other)
Responsible Party: Principal Investigator, Jorge Pereira Machado, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BivalveSarsCov-Protocol; PPA nº 117380 (Registry Identifier: Provisional Patent Application (PPA) by Porto University, Portugal)
Record Dates: First submitted 2021-08-03; First posted 2021-09-23 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus Infections; Coronavirus Sars-Associated; SARS (Severe Acute Respiratory Syndrome); COVID-19
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; COVID-19 | interventions — Fluid Therapy; Fertilization; Infectious Disease Incubation Period; Refrigeration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccinated (Experimental): Subjects that received a vaccine against COVID-19 lineage virus
  Interventions: Biological: Marine liquid and fluids; Biological: Impregnation; Biological: Incubation; Biological: Manipulation; Biological: Refrigeration
- Non-vaccinated (Experimental): Subjects that did not receive a vaccine against COVID-19 lineage virus
  Interventions: Biological: Marine liquid and fluids; Biological: Impregnation; Biological: Incubation; Biological: Manipulation; Biological: Refrigeration
- Infected (Experimental): Subjects that are infected with a COVID-19 lineage virus
  Interventions: Biological: Marine liquid and fluids; Biological: Impregnation; Biological: Incubation; Biological: Manipulation; Biological: Refrigeration

INTERVENTIONS:
Biological: Marine liquid and fluids — Marine liquid and fluids extracted from freshwater bivalve of A. cygnea (under very specific conditions)
Biological: Impregnation — SARS / COVID-19 fluid/liquid - impregnation
Biological: Incubation — SARS / COVID-19 fluid-bivalve-incubation
Biological: Manipulation — Bivalve Manipulation - Stress inducing
Biological: Refrigeration — Refrigerated fluid to check for maintained response

SUMMARY:
The present work proposes to find if a bio-active composite in the hemolymph or plasma of the freshwater bivalve Anodonta cygnea is able to offer immunity and specificity for meliorating the major symptoms in human SARS and COVID-19 lineage infection. The Methodology concerns in silico procedures using organic fluids from 54 bivalves (in very specific conditions) to evaluate their therapeutic effects in 6 voluntary SARS and COVID-19 infected persons with an integrative diagnosis by a computational Mora®Nova apparatus to access the basal and experimental human physiological parameters.

DETAILED DESCRIPTION:
A deep and consistent study will be developed with an increase in the human sampling for better understanding the intervention efficacy of this intelligence medicine integrator, the Mora® Nova method. These in silico experiments when associated with the bioresonance frequencies from stimulated hemolymph compounds of the freshwater bivalve A. cygnea, may lead us to expect high plasticity and immunological potential.

Obviously, additional in vitro studies in future, with adequate culture cell lineages in different conditions and with bioresonance treatment by Mora® Nova method, should also be accomplished with hemolymph/plasma interference to confirm the pertinence, and the real efficacy on SARS / COVID-19 infection as well as to clarify the respective biological mechanisms.

In addition, to analyze and evaluate any specific bioactive compound from the induced hemolymph condition needs molecular experiments which can give deep structural information concerning any efficient molecule against the SARS / COVID-19 virus lineage and respective mutants. Effectively, according to current scientific opinion, the virus mutation phenomenon leads to great and problematic difficulty for maintaining the collective and human global immunization. In this case, the present Mora methodology offers a very functional, dynamic, and efficient process when combined with a biological model, as the bivalve A. cygnea, with high plasticity and eventual molecular reconstructive adaptation. This Mora procedure can extend to other immune-depressive diseases namely cancer, rheumatoid arthritis, and neurodegenerative diseases combining with respective stimulated bivalve fluids. It suggests opening a promising future perspective when applied to large human sampling as well as with in vitro cellular assays.

In addition, to explore this research with in vitro cell cultures and to do the characterization and the effects from bio-compounds on similar diseases is our close objective.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with normal physiological state or any kind of comorbidity

Exclusion Criteria:

* Subjects in highly critical health state

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Pulmonary system | T0 - Day 1 - Baseline
  Voll Electromagnetic conductance reading (Hz) on pulmonary system biopoints
Pulmonary system change | T1 - Day 1 - After in silico human virus infestation
  Voll Electromagnetic conductance reading (Hz) on pulmonary system biopoints
Pulmonary system change | T2 - Day 1 - After adding the interface of the original fluid
  Voll Electromagnetic conductance reading (Hz) on pulmonary system biopoints
Pulmonary system change | T3 - Day 1 - After adding the interface of virus impregnated fluid
  Voll Electromagnetic conductance reading (Hz) on pulmonary system biopoints
Pulmonary system change | T4 - Day 3 - After adding the interface of virus incubated fluid during 48 hours
  Voll Electromagnetic conductance reading (Hz) on pulmonary system biopoints
Cardiac system | T0 - Day 1 - Baseline
  Voll Electromagnetic conductance reading (Hz) on cardiac system biopoints
Cardiac system change | T1 - Day 1 - After in silico human virus infestation
  Voll Electromagnetic conductance reading (Hz) on cardiac system biopoints
Cardiac system change | T2 - Day 1 - After adding the interface of the original fluid
  Voll Electromagnetic conductance reading (Hz) on cardiac system biopoints
Cardiac system change | T3 - Day 1 - After adding the interface of virus impregnated fluid
  Voll Electromagnetic conductance reading (Hz) on cardiac system biopoints
Cardiac system change | T4 - Day 3 - After adding the interface of virus incubated fluid during 48 hours
  Voll Electromagnetic conductance reading (Hz) on cardiac system biopoints
Immunologic system | T0 - Day 1 - Baseline
  Voll Electromagnetic conductance reading (Hz) on immunologic system biopoints
Immunologic system change | T1 - Day 1 - After in silico human virus infestation
  Voll Electromagnetic conductance reading (Hz) on immunologic system biopoints
Immunologic system change | T2 - Day 1 - After adding the interface of the original fluid
  Voll Electromagnetic conductance reading (Hz) on immunologic system biopoints
Immunologic system change | T3 - Day 1 - After adding the interface of virus impregnated fluid
  Voll Electromagnetic conductance reading (Hz) on immunologic system biopoints
Immunologic system change | T4 - Day 3 - After adding the interface of virus incubated fluid during 48 hours
  Voll Electromagnetic conductance reading (Hz) on immunologic system biopoints

SECONDARY OUTCOMES:
Gastrointestinal system | T0 - Day 1 - Baseline
  Voll Electromagnetic conductance reading (Hz) on gastrointestinal system biopoints
Gastrointestinal system Change | T1 - Day 1 - After in silico human virus infestation
  Voll Electromagnetic conductance reading (Hz) on gastrointestinal system biopoints
Gastrointestinal system Change | T2 - Day 1 - After adding the interface of the original fluid
  Voll Electromagnetic conductance reading (Hz) on gastrointestinal system biopoints
Gastrointestinal system Change | T3 - Day 1 - After adding the interface of virus impregnated fluid
  Voll Electromagnetic conductance reading (Hz) on gastrointestinal system biopoints
Gastrointestinal system Change | T4 - Day 3 - After adding the interface of virus incubated fluid during 48 hours
  Voll Electromagnetic conductance reading (Hz) on gastrointestinal system biopoints
Nervous system | T0 - Day 1 - Baseline
  Voll Electromagnetic conductance reading (Hz) on nervous system biopoints
Nervous system change | T1 - Day 1 - After in silico human virus infestation
  Voll Electromagnetic conductance reading (Hz) on nervous system biopoints
Nervous system change | T2 - Day 1 - After adding the interface of the original fluid
  Voll Electromagnetic conductance reading (Hz) on nervous system biopoints
Nervous system change | T3 - Day 1 - After adding the interface of virus impregnated fluid
  Voll Electromagnetic conductance reading (Hz) on nervous system biopoints
Nervous system change | T4 - Day 3 - After adding the interface of virus incubated fluid during 48 hours
  Voll Electromagnetic conductance reading (Hz) on nervous system biopoints
Endocrine system | T0 - Day 1 - Baseline
  Voll Electromagnetic conductance reading (Hz) on endocrine system biopoints
Endocrine system change | T1 - Day 1 - After in silico human virus infestation
  Voll Electromagnetic conductance reading (Hz) on endocrine system biopoints
Endocrine system change | T2 - Day 1 - After adding the interface of the original fluid
  Voll Electromagnetic conductance reading (Hz) on endocrine system biopoints
Endocrine system change | T3 - Day 1 - After adding the interface of virus impregnated fluid
  Voll Electromagnetic conductance reading (Hz) on endocrine system biopoints
Endocrine system change | T4 - Day 3 - After adding the interface of virus incubated fluid during 48 hours
  Voll Electromagnetic conductance reading (Hz) on endocrine system biopoints

CONTACTS AND LOCATIONS:
Overall Officials: Jorge P Machado, PhD, Study Director — ICBAS - Instituto de Ciências Biomédicas Abel Salazar
Locations (2):
- Portugal (2):
  - Instituto Politécnico de Bragança, Bragança
  - ICBAS - University of Porto, Porto

REFERENCES:
- [Background] Antunes F, Hinzmann M, Lopes-Lima M, Machado J, Martins da Costa P. Association between environmental microbiota and indigenous bacteria found in hemolymph, extrapallial fluid and mucus of Anodonta cygnea (Linnaeus, 1758). Microb Ecol. 2010 Aug;60(2):304-9. doi: 10.1007/s00248-010-9649-y. Epub 2010 Mar 27. PMID 20349058
- [Background] Le Bert N, Tan AT, Kunasegaran K, Tham CYL, Hafezi M, Chia A, Chng MHY, Lin M, Tan N, Linster M, Chia WN, Chen MI, Wang LF, Ooi EE, Kalimuddin S, Tambyah PA, Low JG, Tan YJ, Bertoletti A. SARS-CoV-2-specific T cell immunity in cases of COVID-19 and SARS, and uninfected controls. Nature. 2020 Aug;584(7821):457-462. doi: 10.1038/s41586-020-2550-z. Epub 2020 Jul 15. PMID 32668444
- [Background] Allam B, Raftos D. Immune responses to infectious diseases in bivalves. J Invertebr Pathol. 2015 Oct;131:121-36. doi: 10.1016/j.jip.2015.05.005. Epub 2015 May 21. PMID 26003824
- [Background] Green TJ, Speck P. Antiviral Defense and Innate Immune Memory in the Oyster. Viruses. 2018 Mar 16;10(3):133. doi: 10.3390/v10030133. PMID 29547519
- [Background] Guo L, Ren L, Yang S, Xiao M, Chang D, Yang F, Dela Cruz CS, Wang Y, Wu C, Xiao Y, Zhang L, Han L, Dang S, Xu Y, Yang QW, Xu SY, Zhu HD, Xu YC, Jin Q, Sharma L, Wang L, Wang J. Profiling Early Humoral Response to Diagnose Novel Coronavirus Disease (COVID-19). Clin Infect Dis. 2020 Jul 28;71(15):778-785. doi: 10.1093/cid/ciaa310. PMID 32198501
- [Background] Sousa H, Hinzmann M. Review: Antibacterial components of the Bivalve's immune system and the potential of freshwater bivalves as a source of new antibacterial compounds. Fish Shellfish Immunol. 2020 Mar;98:971-980. doi: 10.1016/j.fsi.2019.10.062. Epub 2019 Oct 30. PMID 31676427